CLINICAL TRIAL: NCT02819583
Title: Study Evaluating the Efficacy and Safety of PCAR-019 in CD19 Positive Relapsed or Refractory Leukemia and Lymphoma
Brief Title: CAR-T Cell Immunotherapy in CD19 Positive Relapsed or Refractory Leukemia and Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: The First People's Hospital of Hefei (Other); Hefei Binhu Hospital (Other); Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-019-001
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Acute Lymphocytic Leukemia; Chronic Lymphocytic Leukemia; Follicular Lymphoma; Mantle Cell Lymphoma; B-cell Prolymphocytic Leukemia; Diffuse Large Cell Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Prolymphocytic, B-Cell; Lymphoma, Large B-Cell, Diffuse | interventions — Immunotherapy, Adoptive; Sensitivity and Specificity; Antigens, CD19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PCAR-019 (Experimental): Enrolled patients will receive PCAR-019 with a novel specific chimeric antigen receptor targeting CD19 antigen by infusion.
  Interventions: Biological: PCAR-019 (anti-CD19 CAR-T cells)

INTERVENTIONS:
Biological: PCAR-019 (anti-CD19 CAR-T cells)
  Other Names: chimeric antigen receptor T cells with specificity for CD19

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of CAR-T cell immunotherapy in patients with CD19 positive relapsed or refractory Leukemia and Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

Male and female subjects with CD19+ B cell malignancies in patients with no available curative treatment options (such as autologous or allogeneic SCT) who have limited prognosis (several months to < 2 year survival) with currently available therapies will be enrolled:

1. Eligible diseases: Acute lymphocytic leukemia (ALL), Chronic lymphocytic leukemia (CLL), Follicular lymphoma, Mantle cell lymphoma, B-cell prolymphocytic leukemia, and diffuse large cell lymphoma, previously identified as CD19+.
2. Patients 18 years of age or older, and must have a life expectancy > 12 weeks.
3. Eastern cooperative oncology group (ECOG) performance status of 0-2 or karnofsky performance status (KPS) score is higher than 60.
4. Adequate venous access for apheresis or venous sampling, and no other contraindications for leukapheresis.
5. Females of child-bearing potential must have a negative pregnancy test and all subjects must agree to use an effective method of contraception for up to two weeks after the last infusion of CAR T cells.
6. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements: White blood cell count (WBC) ≥ 2500c/ml, Platelets ≥ 50×10^9/L, Hb ≥ 9.0g/dL, lymphocyte (LY) ≥ 0.7×10^9/L, LY% ≥ 15%, Alb ≥ 2.8g/dL, serum lipase and amylase < 1.5×upper limit of normal, serum creatinine ≤ 2.5mg/dL, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5×upper limit of normal, serum total bilirubin ≤ 2.0mg/dL. These tests must be conducted within 7 days prior to registration.
7. Ability to give informed consent.

Exclusion Criteria:

1. The transduction efficiency of the T cells is less than 30% or the amplification of the T cells via artificial antigen presenting cell (aAPC) stimulation is less than 5 times.
2. Pregnant or nursing women may not participate.
3. Active HIV, hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at the time of screening.
4. Serious illness or medical condition which would not permit the patient to be managed according to the protocol, including active uncontrolled infection, major cardiovascular, coagulation disorders, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive/restrictive pulmonary disease, or psychiatric or emotional disorders.
5. History of severe immediate hypersensitivity to any of the agents including cyclophosphamide, fludarabine, or aldesleukin.
6. Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary.
7. Previously treatment with any gene therapy products.
8. The existence of unstable or active ulcers or gastrointestinal bleeding.
9. Patients need anticoagulant therapy (such as warfarin or heparin).
10. Patients need long-term antiplatelet therapy (aspirin at a dose > 300mg/d; clopidogrel at a dose > 75mg/d).
11. Patients using fludarabine or cladribine chemotherapy within 3 months prior to leukapheresis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Phase I: Adverse events attributed to the administration of the anti-CD19 CAR-T cells | 2 years

SECONDARY OUTCOMES:
Phase II: Objective Response Rate | Safety follow-up is 100 days from last CAR-T infusion.

CONTACTS AND LOCATIONS:
Locations (1):
- PersonGen BioTherapeutics (Suzhou) Co., Ltd., Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes